CLINICAL TRIAL: NCT03049644
Title: Management of Chronic Lower Back Pain: A Randomized Controlled Trial Comparing Mechanical Diagnosis and Treatment to Manual Therapy Utilizing a Point of Care Methodology
Brief Title: A Trial Comparing Mechanical Diagnosis and Treatment to Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Dougherty, DC, Chief of Chiropractic/Residency Director, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 977015
Record Dates: First submitted 2017-02-01; First posted 2017-02-10 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Chronic Lower Back Pain
Keywords: chronic lower back pain; Manual Therapy; Mechanical Diagnosis and Treatment
MeSH Terms: interventions — Therapeutics; Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical Diagnosis and Therapy (Active Comparator): Mechanical diagnosis refers to the classification based on examination of posture and range of motion of the spine, associated with the assessment of subjective symptomatic responses.
  Interventions: Procedure: Mechanical Diagnosis and Therapy
- Manual Therapy (Active Comparator): Manual therapy (MT) is a broad term encompassing many techniques which attempt to affect possible pain contributors such as joints, tendons, ligaments, and muscles, typically using the therapist's hands but may also utilize a tool or instrument in the case of some soft tissue mobilization therapies as well as low force instrument assisted spinal manipulation therapy.
  Interventions: Procedure: Manual Therapy

INTERVENTIONS:
Procedure: Mechanical Diagnosis and Therapy — Identification of directional preference.
  Other Names: McKenzie
  Arms: Mechanical Diagnosis and Therapy
Procedure: Manual Therapy — Mechanically based treatment based on taking joint to end range and thrusting or soft tissue manipulation.
  Other Names: Spinal Manipulative therapy
  Arms: Manual Therapy

SUMMARY:
Mechanical diagnosis and treatment (MDT) and Manual Therapy (MT) have both demonstrated efficacy in the management of CLBP. The use of a Point of Care (POC) design in this study will allow for comparison of these two treatment modalities in a clinical setting. The purpose of this study is to demonstrate the feasibility of recruiting, enrolling and collecting outcome data on CLBP patients utilizing the POC methodology.

DETAILED DESCRIPTION:
20 new patients entering the chiropractic clinic who meet inclusion criteria including demonstrating a directional preference upon physical examination during their initial evaluation will be recruited. Patients will be queried as to interest and those interested will be consented. Patients will then be randomized utilizing a computer generated randomization chart to receive either MDT or MT delivered in a pragmatic manner. Outcomes will include: Pain (PEG), Quality of Life (PROMIS Global Health Survey (GHS)), psychosocial questions and Self Efficacy (2 Question). Outcomes will be collected at baseline, 4 weeks and 8 weeks post baseline.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Lower back pain (CLBP) (>12 weeks)
* Veteran
* At least 18 years of age
* Directional preference on physical examination

Exclusion Criteria:

* Non Veteran
* >89 years of age
* Non Mechanical Cause of LBP
* Unable to identify directional preference on physical examination
* Contraindications to manual therapy (cauda equina syndrome, spinal neoplasia or metastatic disease, destructive joint pathology such as rheumatoid arthritis, bowel/bladder dysfunction (associated with the back pain), peripheral neuropathy or progressive lumbosacral radiculopathy, progressive myelopathy or neurogenic claudication or any absolute contraindications to MT such as acute fracture of the lumbar spine)
* Open Worker's compensation case

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
PROMIS Global Health Scale (GHS) | baseline, 4 week and 8 week (assessing change from baseline to 4 weeks and 8 weeks)
  Change in Quality of Life Measure

SECONDARY OUTCOMES:
PEG (Pain/enjoyment of life/general activity) | baseline, 4 week and 8 week (assessing change from baseline to 4 weeks and 8 weeks)
  Change in Pain
Fear Avoidance | baseline, 4 week and 8 week (assessing change from baseline to 4 weeks and 8 weeks)
  It's not really safe for a person with my back problem to be physically active (1-5 scale)
Catastrophizing | baseline, 4 week and 8 week (assessing change from baseline to 4 weeks and 8 weeks)
  I feel that my back pain is terrible and it's never going to get any better (1-5 scale)
Behavioral Disengagement | baseline, 4 week and 8 week (assessing change from baseline to 4 weeks and 8 weeks)
  Due to my chronic back pain, I no longer engage in activities that are enjoyable and pleasant (1-5 scale_

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Dougherty, DC, Principal Investigator — Canandaigua VA Medical Center
Locations (1):
- Rochester Outpatient Clinic (ROPC) of the Canandaigua VA Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will publish results of study in a journal as a pilot study.